CLINICAL TRIAL: NCT05701293
Title: A ProspeCtive mUlticenteR Investigation on RENzar Stent Safety and Efficacy in the Treatment of Patients With Femoro-popliteal Disease in Tuscany (CURRENT Registry)
Acronym: CURRENT
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Gianmarco de Donato, Professor, University of Siena
Other Study IDs: Current01
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; chronic limb threatening ischemia; endovascular treatment
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LEAD patients undergoing endovascular treatment with implantation of Renzan stent
  Interventions: Procedure: Endovascular implantation of Renzan Stent

INTERVENTIONS:
Procedure: Endovascular implantation of Renzan Stent — Endovascular treatment of LEAD patients with Renzan Stent

SUMMARY:
CURRENT Registry is a physician-initiated prospective, multicenter, post-market, single-arm study with a plan to include approximately 100 patients eligible to be treated with RenzanTM Peripheral Stent System.

DETAILED DESCRIPTION:
In the last years, most of the technical evolution of materials dedicated to the treatment of femoropopliteal disease has been focused on drug-eluting technologies. However, in very complex lesions drug-coated balloons seems to be less efficient, leading to a high rate of bailout stenting with bare metal stents. Drug-eluting stents have raised expectation, providing structural scaffolding of the artery and active pharmacological treatment of the target lesion. Available evidence from the literature does not always seem to support this hypothesis.

Still, a lot of rumours have been generated on the potential local and systemic toxicity of paclitaxel.

As a consequence, in complex lesion rather than Drug Coated Balloon and Drug Eluting Stent it seems that there is need of a modern generation of nitinol stents with high Radial Resistive Force, low chronic outward forces and high fracture resistance.

The device under investigation is the Renzan™ Peripheral Stent System from Terumo MicroVention Inc. (35 Enterprise, Aliso Viejo, California 92656, USA) .

The System consists of a self-expanding nitinol stent pre-mounted on the distal portion of a rapid exchange (RX) delivery catheter. The stent is made of a nickel-titanium alloy with radiopaque markers on each end of the stent. The nitinol stent is constructed from 2 layers of tubular braided nitinol wire mesh. The outer layer consists of nitinol wire braided into a closed cell structure with flared ends. The inner layer consists of nitinol wire braided into a closed cell structure with micro sized pores. The delivery catheter has a rapid exchange port designed to allow coaxial passage of a 0.46mm (0.018") or smaller guide wire in diameter. The stent is capable of being recaptured when a minimum of 20mm of stent length remains inside the catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Subject must provide written informed consent prior to the treatment of the target lesion.
3. Subject must be willing to comply with the specified follow-up evaluation schedule.
4. Subject with Rutherford-Becker clinical classification category 2 to 5, with a resting ankle-brachial index (ABI) ≤ 0.9.
5. Common femoral, superficial femoral and/or popliteal artery lesion with > 50% stenosis or total occlusion.
6. Stenotic or occluded lesion(s) within the same vessel with no length limits.
7. De novo or restenotic/occluded lesion(s) including in-stent restenosis, with reference vessel diameter (RVD) ≥ 4.0 mm and ≤ 8.0 mm by visual assessment and no length limits.
8. Multiple RENZAN stents could be deployed with a mandatory overlap of 0.5-1 cm.
9. A patent inflow artery free from the significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of ipsilateral iliac lesions); Successful ipsilateral iliac artery treatment is defined as the attainment of residual diameter stenosis ≤30%, either with PTA or stenting.
10. The target lesion(s) can be successfully crossed with a guide wire and dilated up to 1:1 to the proposed stent to be implanted (as per the operator's assessment).
11. At least one patent native outflow artery (anterior or posterior tibial or peroneal), free from significant (≥50%) stenosis (as confirmed by angiography), that has not previously been revascularized. The remaining outflow arteries requiring treatment during the same procedure may be treated

Exclusion Criteria:

1. Subject has Rutherford-Becker classification category 6.
2. Treatment of lesions requiring the use of adjunctive debulking devices.
3. Use of drug-eluting balloon or stent
4. Inadequate vessel preparation not achieving a diameter of 1:1 to the stent to be implanted (with ≤20% residual stenosis, as per operator's assessment).
5. Concomitant use of different stent platforms
6. Any significant vessel tortuosity or other parameters prohibiting access to the lesion and/or preventing the stent delivery.
7. Subject with coronary intervention performed less than 90 days prior to or planned within 30 days after the treatment of the target lesion.
8. Known allergies or intolerance to nitinol (nickel titanium).
9. Any contraindication or known unresponsiveness to dual antiplatelet therapy (DAPT) or anticoagulation therapy.
10. Presence of acute thrombus prior to crossing the lesion.
11. Thrombolysis of the target vessel within 72 hours prior to the index procedure
12. Thrombophlebitis or deep venous thrombus, within the previous 30 days.
13. Subject receiving dialysis within the previous 30 days.
14. Stroke within the previous 90 days.
15. Subject is pregnant or of childbearing potential
16. Subject has a life expectancy of less than 1 year.
17. Subject is participating in an investigational study that has not reached the primary endpoint at the time of study screening.
18. Only one patent outflow artery, with significant stenosis (≥50%) (as confirmed by angiography)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Lower Extremity Artery disease needing for endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety endpoint [composite] | 30 days after procedure
  Death + target lesion revascularization (TLR) + Major Amputation (above the ankle)
Primary Efficacy endpoint | 12 months
  Primary patency of the artery at 12 months, defined as no evidence of occlusion within the originally treated lesion based on Color Flow Doppler ultrasound in the absence of target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Device Success | Intraoperative
  Successful device deployment according to Instruction For Use.
Technical Success | Intraoperative
  Achievement of a final target lesion residual diameter stenosis of <30% based on angiography.
Procedural Success | Intraoperative
  Technical and device success without procedural complication.
Any death | 1, 6, 12 24 and 36 months
  Cardiovascular death and non-cardiovascular death
Clinically-driven Target Lesion Revascularization (CD-TLR) | 1, 6, 12 24 and 36 months
  Any TLR associated with deterioration of patient's Rutherford category and/or increase in size of pre-existing ischemic wounds and/or occurrence of new wounds.
Patency of Target lesion | 1, 6, 12 24 and 36 months
  Defined as no evidence of restenosis or occlusion within the originally treated lesion based on a Color Flow Doppler ultrasound in the absence of target lesion revascularization (TLR). Occlusion and restenosis were defined as no color flow or an increase in peak systolic velocity ratio (PSVR) of ≥ 2.4 when compared to the proximal normal segment, respectively.
Limb Ischemia Improvement | 1, 6, 12 24 and 36 months
  Improvement in the Rutherford-Becker Clinical Improvement Scale of greater than or equal to 1.
  -Rutherford-Becker Classification: 0 Asymptomatic
  1. Mild claudication
  2. Moderate claudication
  3. Severe claudication
  4. Ischemic rest pain
  5. Minor tissue loss
  6. Major tissue loss
MAE (Major Adverse Event) | 1, 6, 12 24 and 36 months
  a composite rate of:
  * cardiovascular death
  * procedure-related arterial rupture
  * acute limb ischemia
  * stent thrombosis
  * clinically apparent distal embolization
  * target limb amputation
  * procedure-related bleeding event requiring transfusion
Index Limb Amputation | 1, 6, 12 24 and 36 months
  Amputation above the ankle.
Stent deployment performance evaluation | Intraoperative
  Operators feedback on: Pushability/Trackability, Deployment, Visibility and Precise Placement
  -High, Moderate and Low

CONTACTS AND LOCATIONS:
Locations (1):
- University of Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH; GVG Writing Group. Global vascular guidelines on the management of chronic limb-threatening ischemia. J Vasc Surg. 2019 Jun;69(6S):3S-125S.e40. doi: 10.1016/j.jvs.2019.02.016. Epub 2019 May 28. PMID 31159978